CLINICAL TRIAL: NCT02395887
Title: Postural Balance and Stability Among Patients With Cervical and Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, shay shabat, Prof. Shay Shabat, Meir Medical Center
Other Study IDs: MeirMc0297-14CTIL
Record Dates: First submitted 2015-03-04; First posted 2015-03-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Spinal Stenosis; Back Pain
Keywords: Spinal stenosis; Spinal decompression; Postural balance; Neurogenic claudication
MeSH Terms: conditions — Spinal Stenosis; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervational: Patients with back or neck pain who are a candidates for operational intervention.
- Control: Men or women who haven't seek for spine surgery consultation.

SUMMARY:
High percentage of chronic back pain is due to spinal stenosis. The clinical picture is of 'neurogenic claudication' which effects postural balance and stability. If conservative treatment fail to improve symptoms, an invasive treatment which includes spinal decompression can be done.

The research is an observational prospective one, pre and post operational intervention. The aim is to examine whether an operational intervention improves quality of life, pain, postural balance an stability among patients.

It's important to clarify, that although there is operational intervention, the research is observational. The decision weather to operate or not, is not a part of the research. The investigators assume that since there is a population that independently going through an operation, the investigators can observe this population and evaluate different aspects of the operation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from back or neck pain
* Patients that are candidates for operational intervention

Exclusion Criteria:

* Pregnant women
* Patients who had a spinal operation in the past.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients, men and women above 18, which suffer from back or neck pain and are candidates for an operational intervention.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Dynamic postural balance tests | 6 months
Static postural balance tests | 6 months

SECONDARY OUTCOMES:
Pain and quality of life questionnaires | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shay Shabat, MD, Principal Investigator — Meir Medical Center